CLINICAL TRIAL: NCT03816969
Title: A Prospective Randomized Comparative Study Between the Self-pressurized Air-Q With Blocker and Air-Q Blocker in Low Risk Female Patients Undergoing Ambulatory Surgery
Brief Title: Self-pressurized Air-Q With Blocker and Air-Q Blocker in Low Risk Female Patients Undergoing Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N 1- 2018/Ms
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Ambulatory Surgery
Keywords: Self-pressurized Air Q

STUDY DESIGN:
Intervention Model Description: It has a drain tube through which a suction tube is passed like the Air-QILA blocker, and Instead of the pilot balloon and inflating cuff, the air-Q SP with blocker incorporates a self-regulating periglottic cuff at the end of this tube, a communication orifice at the junction of the peri-glottic cuff and the airway tube. This communication between two spaces enables the cuff to dynamically regulate intra-cuff pressure depending on airway pressure. This distinguishing feature of the air-Q SP may result in reduced risk for airway morbidities related to cuff hyperinflation.
Who Masked: Participant, Investigator
Masking Description: An online randomization program (http://www.randomizer.org) will be used to generate random list and to allocate patients into the study groups. Random allocation numbers will be concealed in opaque closed envelops. The patient and investigator assessing study outcomes will all be blinded to the study groups allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-pressurized air-Q with blocker (Active Comparator): Self-pressurized air-Q with blocker has a greater seal pressure compared to Air-Q blocker, easier and faster in insertion and has less morbidity and complications while and after insertion
  Interventions: Device: Self-pressurized air-Q with blocker
- Air-Q ILA blocker (Active Comparator): It has a drain tube through which a suction tube is passed
  Interventions: Device: Air-Q ILA blocker

INTERVENTIONS:
Device: Self-pressurized air-Q with blocker — It has a drain tube through which a suction tube is passed like the Air-QILA blocker, and Instead of the pilot balloon and inflating cuff, the air-Q SP with blocker incorporates a self-regulating periglottic cuff at the end of this tube , a communication orifice at the junction of the peri-glottic cuff and the airway tube.
  This communication between two spaces enables the cuff to dynamically regulate intra-cuff pressure depending on airway pressure. This distinguishing feature of the air-Q SP may result in reduced risk for airway morbidities related to cuff hyperinflation
  Arms: Self-pressurized air-Q with blocker
Device: Air-Q ILA blocker — A good seal will provide good ventilation, will guarantee the desired depth of anesthesia at lower gas flows and with lesser leaks to the esophagus, it will not cause rise in intragastric pressure thus preventing regurgitation However, When the cuff pressure is more than the mucosal perfusion pressure, it is likely to either cause postoperative pharyngo-laryngeal symptoms (sore throat, dysphagia, dysphonia) or cause local mucosal trauma and nerve injuries
  Arms: Air-Q ILA blocker

SUMMARY:
In this study investigators shall compare between the two types of air-Q 's; the Air-Q ILA blocker and the Air-Q SP with blocker , regarding good sealing and oropharyngeal leak pressure

DETAILED DESCRIPTION:
The Air-Q family has introduced many improved designs, among which the Air- Q blocker intubating laryngeal airway (Air-Q ILA blocker) in 2011. It has all the previously mentioned advantages, and in addition, a new, built-in, soft guide channel that accepts regular Nasal Gastric (NG) tubes to suction or optional Blocker Tubes for accessing the posterior pharynx and managing the esophagus. investigators can suction the pharynx or suction, vent and block the upper esophagus. Ever since the idea of SAD has launched and applying an optimum intra-cuff pressure that maintains enough sealing and at the same time not injurious to the oropharyngeal mucosa concerns anesthesiologists A good seal will provide good ventilation, will guarantee the desired depth of anesthesia at lower gas flows and with lesser leaks to the esophagus, it will not cause rise in intragastric pressure thus preventing regurgitation However When the cuff pressure is more than the mucosal perfusion pressure, it is likely to either cause postoperative pharyngo-laryngeal symptoms (sore throat, dysphagia, dysphonia) or cause local mucosal trauma and nerve injuries Therefore, in 2013 another improvised design of the Air-Q family has evolved, a Self-pressurized Air Q (air-Q SP) with blocker) . It has a drain tube through which a suction tube is passed like the Air-QILA blocker , And Instead of the pilot balloon and inflating cuff, the air-Q SP with blocker incorporates a self-regulating periglottic cuff at the end of this tube, a communication orifice at the junction of the peri-glottic cuff and the airway tube. This communication between two spaces enables the cuff to dynamically regulate intra-cuff pressure depending on airway pressure. This distinguishing feature of the air-Q SP may result in reduced risk for airway morbidities related to cuff hyperinflation. In this study investigators shall compare between the two types of air-Q 's; the Air-Q ILA blocker and the Air-Q SP with blocker , regarding good sealing and oropharyngeal leak pressure

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between the age group of 18 and 50 years.
2. Patients of American Society of Anaesthesiologists (ASA) class I and II.
3. Patients with Ganzouri airway score less than 4.

Exclusion Criteria:

1. ASA III - V patients.
2. Airway score ≥ 4 according to El-Ganzouri Airway Scoring System.
3. Patients with any oropharyngeal pathology.
4. Patients known to have risk of gastric aspiration, gastro-esophageal reflux disease, hiatus hernia or previous upper gastrointestinal tract surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 10 Minutes after initial assessment
  The Oropharyngeal leak pressure after insertion and fixation of the device

SECONDARY OUTCOMES:
Insertion time | 10 Minutes
  time of insertion
Complications associated | 24 hours
  Hypoxemia (SpO2 <90%), intra and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Press